CLINICAL TRIAL: NCT06340945
Title: The Clinical Outcomes and Artificial Intelligence Prediction Model of Ultrasound-guided Thermal Ablation for the Treatment of Benign Thyroid Nodules：A Multicenter Prospective Study
Brief Title: The Outcomes of Ultrasound-guided Thermal Ablation for Benign Thyroid Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-kun Luo, Director, Head of Department of Ultrasound, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S2023-761-01
Record Dates: First submitted 2024-03-16; First posted 2024-04-02 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Nodules
MeSH Terms: conditions — Thyroid Nodule | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound-guided thermal ablation (Experimental)
  Interventions: Procedure: ultrasound-guided thermal ablation

INTERVENTIONS:
Procedure: ultrasound-guided thermal ablation — microwave ablation, radio frequency ablation, laser ablation

SUMMARY:
1. To evaluate the clinical outcomes of ultrasound-guided thermal ablationfor the treatment of benign thyroid nodules;
2. To develop and validate a artificial intelligence model to predict the outcomes of ultrasound-guided thermal ablation in the treatment of benign thyroid nodules

ELIGIBILITY:
Inclusion Criteria:

* [1]confirmation of benign nodule status on two separate fine- needle aspiration (FNA) or core-needle biopsy (CNB) [2]no suspicious malignant features on ultrasound examination [3]report of cosmetic and/ or symptomatic problems or concern of nodules growing rapidly or malignant transformation [4]refusal or ineligibility for surgery [5]follow-up time ≥6months

Exclusion Criteria:

1. follicular neoplasm or malignancy findings on biopsy
2. nodules with benign result on biopsy had suspicious of malignancy in US, including marked hypoechoic, ill-defined margins, taller-than-wide shape or microcalcifications
3. patients with cystic nodules
4. patients with contra-lateral vocal cord par- alysis
5. previous radiation to the head and neck
6. ; follow- up time less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
volume reduction rate | through study completion, an average of 6 months
  The volume reduction rate (VRR)was calculated by the equations: VRR=([initial volume-final volume] × 100)/initial volume
rate of nodule regrowth | through study completion, an average of 1 months
  Regrowth was defined as ≥50% volume increase compared to the previously recorded smallest volume during the follow-up

SECONDARY OUTCOMES:
rate of complications | 1 week
  complications after ablation
cosmetic score | through study completion, an average of 6 months
  The cosmetic score was assessed by a physician (1, no palpable mass; 2, no cosmetic problem but palpable mass; 3, a cosmetic problem on swallowing only; and 4, a readily detected cosmetic problem)
symptom score | through study completion, an average of 6 months
  The symptom score was self-measured by patients using a 10-cm visual analogue scale (grade 0-10)
vital volume | through study completion, an average of 6 months
  vital volume was the incompletely treated vital volume which located peripherally
total volume | through study completion, an average of 6 months
  the overall volume of the nodules

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No